CLINICAL TRIAL: NCT00597753
Title: AFX01-12: A Phase 3, Randomized, Active-controlled, Open-label, Multi-center Study of the Safety and Efficacy of Peginesatide for the Maintenance Treatment of Anemia in Hemodialysis Patients Previously Treated With Epoetin Alfa
Brief Title: Safety & Efficacy of Peginesatide for Maintenance Treatment of Anemia in Participants With Chronic Kidney Disease on Hemodialysis
Acronym: EMERALD 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Affymax (Industry)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AFX01-12
Record Dates: First submitted 2008-01-10; First posted 2008-01-18 (Estimated); Results first posted 2012-07-30 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-02

CONDITIONS: Chronic Renal Failure; Chronic Kidney Disease; Anemia
Keywords: anemia; chronic kidney disease; CKD; chronic renal failure; CRF; dialysis; erythropoietin; EPO; erythropoiesis stimulating agent; ESA; Hematide™; hemodialysis; hemoglobin; Hb; Hgb; Omontys; peginesatide; red blood cell; red blood cell production
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic; Anemia | interventions — peginesatide; hematide; Epoetin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Peginesatide (Experimental)
  Interventions: Drug: peginesatide
- Epoetin alfa (Active Comparator)
  Interventions: Drug: Epoetin Alfa

INTERVENTIONS:
Drug: peginesatide — Participants received peginesatide by intravenous injection once every 4 weeks. The starting dose was based on the participant's total weekly epoetin alfa dose during the last week of the Screening Period; the first dose was administered one week after the last epoetin alfa dose. The dose was adjusted to maintain hemoglobin levels in a target range of 10.0-12.0 grams per deciliter (g/dL) and ± 1.5 g/dL from baseline during the Titration and Evaluation Periods, and 10.0-12.0 g/dL during the Long-Term Safety and Efficacy Period.
  Other Names: Omontys; Hematide; AF37702 Injection
  Arms: Peginesatide
Drug: Epoetin Alfa — Participants continued to receive commercially available epoetin alfa by intravenous injection, at the same starting dose and frequency as received during the last week of the Screening Period, with the first study dose of epoetin alfa administered after randomization at Week 0. The dose was adjusted to maintain hemoglobin levels in a target range of 10.0-12.0 g/dL and ± 1.5 g/dL from baseline during the Titration and Evaluation Periods, and 10.0-12.0 g/dL during the Long-Term Safety and Efficacy Period.
  Other Names: Epogen
  Arms: Epoetin alfa

SUMMARY:
The purpose of the study was to evaluate the safety and efficacy of peginesatide in the maintenance treatment of anemia in participants on dialysis.

DETAILED DESCRIPTION:
Anemia associated with chronic kidney disease is due to several factors, primarily the inability of the diseased kidneys to produce adequate amounts of endogenous erythropoietin. Ancillary factors include the shortened lifespan of red blood cells, iron and other nutritional deficiencies, infection, and inflammation. The presence and severity of anemia are related to the duration and extent of kidney failure. Anemia is associated with increased mortality, increased likelihood of hospitalization, reduced cognitive function, and increased left ventricular hypertrophy and heart failure.

Erythropoiesis stimulating agents (ESAs) have been established as a treatment for anemia in chronic renal failure subjects, and have improved the management of anemia over alternatives such as transfusion. Peginesatide is a parenteral formulation developed for the treatment of anemia in patients with chronic kidney disease. Peginesatide binds to and activates the human erythropoietin receptor, and stimulates erythropoiesis in human red cell precursors in a manner similar to other known erythropoiesis-stimulating agents.

Eligible participants were randomized in a 2:1 ratio to peginesatide administered once every 4 weeks or to continued treatment with epoetin alfa administered 1-3 times each week, respectively. Total commitment time for this study was 4 weeks of screening followed by a minimum of 52 weeks of study treatment.

To evaluate the cardiovascular safety of peginesatide, a cardiovascular composite safety endpoint (CSE) was defined for use in prospectively planned analyses which combined cardiovascular safety data from the four Phase 3 peginesatide studies (NCT00598273, NCT00597753, NCT00598442, and NCT00597584). The CSE consisted of six events: death, stroke, myocardial infarction, and serious adverse events of congestive heart failure, unstable angina, and arrhythmia. An independent Event Review Committee (ERC) was used to provide blinded adjudication of potential CSE events.

ELIGIBILITY:
Inclusion Criteria

1. Participants with chronic renal failure on hemodialysis for ≥ 3 months prior to randomization.
2. On intravenous epoetin alfa maintenance therapy continuously prescribed for a minimum of 8 weeks prior to randomization.
3. Four consecutive hemoglobin values with a mean ≥ 10.0 and ≤ 12.0 g/dL during the screening period

Exclusion Criteria

1. Females who are pregnant or breast-feeding.
2. Known intolerance to any erythropoiesis stimulating agent (ESA) or pegylated molecule or to all parenteral iron supplementation products.
3. Known bleeding or coagulation disorder.
4. Known hematologic disease or cause of anemia other than renal disease
5. Poorly controlled hypertension
6. Evidence of active malignancy within one year prior to randomization.
7. Temporary (untunneled) dialysis access catheter.
8. A scheduled kidney transplant
9. A scheduled surgery that may be expected to lead to significant blood loss.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 803 (Actual)
Dates: Start 2007-09; Primary Completion 2009-07 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vice President, Clinical Development, Study Director — Affymax
Locations (80):
- United States (80):
  - Research Facility, Paragould, Arkansas
  - Research Facility, Fairfield, California
  - Research Facility, Granada Hills, California
  - Research Facility, Los Alamitos, California
  - Research Facility, Los Angeles, California
  - Research Facility, Lynwood, California
  - Research Facility, Monterey Park, California
  - Research Facility, Mountain View, California
  - Research Facility, Paramount, California
  - Research Facilities (2), San Diego, California
  - Research Facility, San Dimas, California
  - Research Facility, Whittier, California
  - Research Facility, Denver, Colorado
  - Research Facility, Middlebury, Connecticut
  - Research Facility, Hudson, Florida
  - Research Facility, Ocala, Florida
  - Research Facility, Orlando, Florida
  - Research Facility, Pembroke Pines, Florida
  - Research Facility, Augusta, Georgia
  - Research Facility, Decatur, Georgia
  - Research Facility, Marietta, Georgia
  - Research Facility, Honolulu, Hawaii
  - Research Facility, Boise, Idaho
  - Research Facility, Chicago, Illinois
  - Research Facility, Evergreen Park, Illinois
  - Research Facility, Gurnee, Illinois
  - Research Facility, Peoria, Illinois
  - Research Facility, Evansville, Indiana
  - Research Facility, Wichita, Kansas
  - Research Facility, Lexington, Kentucky
  - Research Facility, Baton Rouge, Louisiana
  - Research Facility, Lafayette, Louisiana
  - Research Facility, New Orleans, Louisiana
  - Research Facility, Shreveport, Louisiana
  - Research Facility, Bethesda, Maryland
  - Research Facility, Rockville, Maryland
  - Research Facility, Fall River, Massachusetts
  - Research Facility, Worcester, Massachusetts
  - Research Facility, Dearborn, Michigan
  - Research Facility, Kalamazoo, Michigan
  - Research Facility, Columbus, Mississippi
  - Research Facility, Tupelo, Mississippi
  - Research Facility, St Louis, Missouri
  - Research Facility, Las Vegas, Nevada
  - Research Facility, Eatontown, New Jersey
  - Research Facility, Brooklyn, New York
  - Research Facility, New York, New York
  - Research Facility, The Bronx, New York
  - Research Facility, Williamsville, New York
  - Research Facility, Yonkers, New York
  - Research Facility, Durham, North Carolina
  - Research Facility, Raleigh, North Carolina
  - Research Facility, Canton, Ohio
  - Research Facility, Cincinnati, Ohio
  - Research Facility, Columbus, Ohio
  - Research Facility, Roseburg, Oregon
  - Research Facility, Allentown, Pennsylvania
  - Research Facility, Philadelphia, Pennsylvania
  - Research Facility, Pittsburgh, Pennsylvania
  - Research Facilities (2), Greenville, South Carolina
  - Research Facility, Sumter, South Carolina
  - Research Facility, Dyersburg, Tennessee
  - Research Facility, Knoxville, Tennessee
  - Research Facility, Nashville, Tennessee
  - Research Facility, Arlington, Texas
  - Research Facility, Fort Worth, Texas
  - Research Facility, Grand Prairie, Texas
  - Research Facilities (2), Houston, Texas
  - Research Facility, Houston, Texas
  - Research Facility, McAllen, Texas
  - Research Facility, San Antonio, Texas
  - Research Facility, Tyler, Texas
  - Research Facility, Alexandria, Virginia
  - Research Facility, Chesapeake, Virginia
  - Research Facility, Fairfax, Virginia
  - Research Facility, Mechanicsville, Virginia
  - Research Facilities (2), Norfolk, Virginia
  - Research Facility, Morgantown, West Virginia
  - Research Facility, Appleton, Wisconsin
  - Research Facility, Oshkosh, Wisconsin

REFERENCES:
- [Result] Fishbane S, Schiller B, Locatelli F, Covic AC, Provenzano R, Wiecek A, Levin NW, Kaplan M, Macdougall IC, Francisco C, Mayo MR, Polu KR, Duliege AM, Besarab A; EMERALD Study Groups. Peginesatide in patients with anemia undergoing hemodialysis. N Engl J Med. 2013 Jan 24;368(4):307-19. doi: 10.1056/NEJMoa1203165. PMID 23343061
- [Derived] Macdougall IC, Provenzano R, Sharma A, Spinowitz BS, Schmidt RJ, Pergola PE, Zabaneh RI, Tong-Starksen S, Mayo MR, Tang H, Polu KR, Duliege AM, Fishbane S; PEARL Study Groups. Peginesatide for anemia in patients with chronic kidney disease not receiving dialysis. N Engl J Med. 2013 Jan 24;368(4):320-32. doi: 10.1056/NEJMoa1203166. PMID 23343062

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Peginesatide | Epoetin Alfa
Started | 532 (Randomization was 2:1 peginesatide to epoetin alfa) | 271
Completed | 366 | 202
Not Completed | 166 | 69
Not completed — Adverse Event | 6 | 2
Not completed — Death | 55 | 29
Not completed — Lack of Efficacy | 2 | 0
Not completed — Lost to Follow-up | 10 | 3
Not completed — Physician Decision | 5 | 1
Not completed — Pregnancy | 1 | 0
Not completed — Withdrawal by Subject | 35 | 12
Not completed — Discontinued Dialysis | 0 | 1
Not completed — Never dosed | 2 | 0
Not completed — Noncompliance | 2 | 1
Not completed — Relocation | 17 | 6
Not completed — Renal transplant | 10 | 3
Not completed — Site closed by sponsor | 19 | 7
Not completed — Site elected to close | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Peginesatide | Epoetin Alfa | Total
Number analyzed (Participants) | 524 | 269 | 793
Age, Categorical [Count of Participants; unit: Participants] — Ten participants were excluded from the full analysis population: 8 participants in the Peginesatide group and 2 participants in the Epoetin Alfa groups. These 10 participants did not receive study medication.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 370 | 190 | 560
    >=65 years | 154 | 79 | 233
Age Continuous [Mean (Standard Deviation); unit: years] | 57.3 (13.96) | 57.5 (13.68) | 57.4 (13.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 231 | 125 | 356
  Male | 293 | 144 | 437

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Hemoglobin Between Baseline and the Evaluation Period
Description: The baseline hemoglobin value is defined as the mean of five hemoglobin values: the four most recent hemoglobin values taken prior to the day of randomization and the value obtained on the day of randomization. The mean hemoglobin during the Evaluation Period for each participant is calculated as the mean of the available hemoglobin values during study Weeks 29 through 36.
Time Frame: Baseline and Weeks 29-36
Population: Full Analysis Population: All randomized participants who received at least one dose of study medication
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Peginesatide | Epoetin Alfa
Number analyzed (Participants) | 524 | 269
g/dL
  Baseline [N=524, 269] | 11.30 (0.523) | 11.32 (0.493)
  Evaluation Period [N=445, 248] | 11.06 (0.932) | 11.25 (0.846)
  Change from Baseline [N=445, 248] | -0.24 (0.956) | -0.09 (0.922)
Statistical Analysis 1: Comparison: Peginesatide vs Epoetin Alfa; The sample size for this study was determined based on a two group evaluation of non-inferiority using the t-distribution (one-sided significance level 0.025) with a non inferiority margin of -1.0 g/dL. A sample size of approximately 750 (peginesatide group of 500 and epoetin alfa group of 250) provided at least 99% power for the evaluation of non-inferiority, assuming an expected treatment difference of 0.0 g/dL and a standard deviation of 1.5 g/dL; Test type: Non-Inferiority or Equivalence — A non-inferiority margin of -1.0 g/dL was used in the primary efficacy assessments. Non-inferiority was established if the lower limit of the two-sided 95% confidence interval for the difference between the means of the primary endpoint (peginesatide minus control ESA) was ≥ -1.0 g/dL; ANOVA; The ANOVA cell means model was used to estimate primary efficacy endpoint within the specified cells formed by the combination of treatment and strata; Least Squares Mean Difference = -0.15, 95% CI 2-sided [-0.30 to -0.01], Standard Error of Mean 0.072

2. Secondary Outcome: Proportion of Participants Who Receive Red Blood Cell (RBC) Transfusions During the Titration and Evaluation Periods
Time Frame: Weeks 0 to 36
Population: Full Analysis Population: All randomized participants who received at least one dose of study medication
Measure: Number; unit: percentage of participants
Arm/Group | Peginesatide | Epoetin Alfa
Number analyzed (Participants) | 524 | 269
percentage of participants | 0.103 | 0.086
Statistical Analysis 1: Comparison: Peginesatide vs Epoetin Alfa; Test type: Superiority or Other; Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.21, 95% CI 2-sided [0.76 to 1.92]

3. Secondary Outcome: Proportion of Participants Whose Mean Hemoglobin Level During the Evaluation Period is Within the Target Range of 10.0 - 12.0 Grams Per Deciliter (g/dL)
Time Frame: Weeks 29 to 36
Population: Full Analysis Population: All randomized participants who received at least one dose of study medication
Measure: Number; unit: percentage of participants
Arm/Group | Peginesatide | Epoetin Alfa
Number analyzed (Participants) | 524 | 269
percentage of participants | 0.630 | 0.717
Statistical Analysis 1: Comparison: Peginesatide vs Epoetin Alfa; Test type: Superiority or Other; Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.88, 95% CI 2-sided [0.79 to 0.97]

ADVERSE EVENTS:
Arm/Group | Peginesatide | Epoetin Alfa
Serious Adverse Events (participants affected / at risk) | 304/524 | 168/269
Other Adverse Events (participants affected / at risk) | 445/524 | 235/269
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Peginesatide (N=524) | Epoetin Alfa (N=269)
Anaemia (Blood and lymphatic system disorders) | 6 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 2
B-lymphocyte abnormalities (Blood and lymphatic system disorders) | 1 | 0
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0
Splenic infarction (Blood and lymphatic system disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 37 | 20
Acute myocardial infarction (Cardiac disorders) | 19 | 9
Myocardial infarction (Cardiac disorders) | 13 | 9
Atrial fibrillation (Cardiac disorders) | 15 | 6
Cardiac arrest (Cardiac disorders) | 16 | 5
Coronary artery disease (Cardiac disorders) | 16 | 5
Angina pectoris (Cardiac disorders) | 12 | 7
Cardio-respiratory arrest (Cardiac disorders) | 11 | 4
Atrial flutter (Cardiac disorders) | 4 | 3
Bradycardia (Cardiac disorders) | 5 | 2
Acute coronary syndrome (Cardiac disorders) | 3 | 3
Angina unstable (Cardiac disorders) | 2 | 2
Cardiomyopathy (Cardiac disorders) | 4 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 3 | 1
Myocardial ischaemia (Cardiac disorders) | 3 | 1
Ventricular tachycardia (Cardiac disorders) | 2 | 2
Ventricular fibrillation (Cardiac disorders) | 3 | 0
Arrhythmia (Cardiac disorders) | 1 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 1 | 1
Coronary artery stenosis (Cardiac disorders) | 1 | 1
Pericardial effusion (Cardiac disorders) | 1 | 1
Supraventricular tachycardia (Cardiac disorders) | 2 | 0
Aortic valve stenosis (Cardiac disorders) | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 0
Bradyarrhythmia (Cardiac disorders) | 1 | 0
Cor pulmonale (Cardiac disorders) | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 1
Cyanosis (Cardiac disorders) | 0 | 1
Electromechanical dissociation (Cardiac disorders) | 1 | 0
Hypertensive cardiomyopathy (Cardiac disorders) | 0 | 1
Hypertensive heart disease (Cardiac disorders) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 1
Mitral valve stenosis (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0
Pericarditis uraemic (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 1 | 0
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 0 | 1
Tuberous sclerosis (Congenital, familial and genetic disorders) | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 1 | 0
Hyperparathyroidism (Endocrine disorders) | 2 | 0
Hyperparathyroidism secondary (Endocrine disorders) | 0 | 1
Hyperparathyroidism tertiary (Endocrine disorders) | 0 | 1
Retinal detachment (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 0
Vitreous haemorrhage (Eye disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 9 | 5
Pancreatitis (Gastrointestinal disorders) | 6 | 3
Abdominal pain (Gastrointestinal disorders) | 4 | 4
Diarrhoea (Gastrointestinal disorders) | 5 | 3
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 | 3
Ascites (Gastrointestinal disorders) | 3 | 3
Diabetic gastroparesis (Gastrointestinal disorders) | 3 | 2
Gastritis (Gastrointestinal disorders) | 2 | 3
Colitis (Gastrointestinal disorders) | 2 | 2
Pancreatitis acute (Gastrointestinal disorders) | 3 | 1
Mallory-Weiss syndrome (Gastrointestinal disorders) | 3 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2
Colitis ischaemic (Gastrointestinal disorders) | 2 | 0
Colonic polyp (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 2
Diverticulum (Gastrointestinal disorders) | 1 | 1
Erosive oesophagitis (Gastrointestinal disorders) | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 1
Ileus (Gastrointestinal disorders) | 2 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 2 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Oesophagitis (Gastrointestinal disorders) | 2 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 1
Duodenitis (Gastrointestinal disorders) | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastritis hypertrophic (Gastrointestinal disorders) | 0 | 1
Gastroduodenitis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 | 0
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 1
Large intestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Odynophagia (Gastrointestinal disorders) | 1 | 0
Oesophageal disorder (Gastrointestinal disorders) | 1 | 0
Oesophageal dysplasia (Gastrointestinal disorders) | 1 | 0
Oesophageal spasm (Gastrointestinal disorders) | 1 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 | 0
Short-bowel syndrome (Gastrointestinal disorders) | 1 | 0
Varices oesophageal (Gastrointestinal disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 13 | 8
Chest pain (General disorders) | 14 | 4
Asthenia (General disorders) | 4 | 5
Pyrexia (General disorders) | 5 | 2
Catheter related complication (General disorders) | 2 | 2
Multi-organ failure (General disorders) | 2 | 1
Oedema peripheral (General disorders) | 2 | 0
Adverse drug reaction (General disorders) | 0 | 1
Catheter site haemorrhage (General disorders) | 0 | 1
Catheter thrombosis (General disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Death (General disorders) | 0 | 1
Drug withdrawal syndrome (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Local swelling (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Sudden cardiac death (General disorders) | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 4 | 1
Cholecystitis acute (Hepatobiliary disorders) | 4 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 2
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 2
Biliary colic (Hepatobiliary disorders) | 1 | 0
Gallbladder disorder (Hepatobiliary disorders) | 0 | 1
Hepatic congestion (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Hepatic mass (Hepatobiliary disorders) | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0
Iodine allergy (Immune system disorders) | 1 | 0
Pneumonia (Infections and infestations) | 37 | 19
Sepsis (Infections and infestations) | 15 | 13
Cellulitis (Infections and infestations) | 15 | 10
Gangrene (Infections and infestations) | 8 | 5
Gastroenteritis (Infections and infestations) | 8 | 5
Staphylococcal bacteraemia (Infections and infestations) | 6 | 7
Urinary tract infection (Infections and infestations) | 11 | 2
Bacteraemia (Infections and infestations) | 5 | 5
Lobar pneumonia (Infections and infestations) | 5 | 5
Septic shock (Infections and infestations) | 6 | 4
Arteriovenous graft site infection (Infections and infestations) | 2 | 7
Osteomyelitis (Infections and infestations) | 4 | 5
Staphylococcal sepsis (Infections and infestations) | 5 | 3
Catheter sepsis (Infections and infestations) | 2 | 5
Bronchitis (Infections and infestations) | 4 | 2
Catheter related infection (Infections and infestations) | 2 | 3
Clostridium difficile colitis (Infections and infestations) | 3 | 2
Staphylococcal infection (Infections and infestations) | 3 | 2
Diverticulitis (Infections and infestations) | 2 | 2
Upper respiratory tract infection (Infections and infestations) | 2 | 2
Abscess limb (Infections and infestations) | 1 | 2
Arteriovenous fistula site infection (Infections and infestations) | 0 | 3
Diabetic foot infection (Infections and infestations) | 2 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 2
Localised infection (Infections and infestations) | 2 | 1
Oesophageal candidiasis (Infections and infestations) | 2 | 1
Appendicitis (Infections and infestations) | 2 | 0
Arthritis bacterial (Infections and infestations) | 1 | 1
Bacterial sepsis (Infections and infestations) | 1 | 1
Catheter bacteraemia (Infections and infestations) | 2 | 0
Device related infection (Infections and infestations) | 1 | 1
Enterocolitis infectious (Infections and infestations) | 2 | 0
Haematoma infection (Infections and infestations) | 2 | 0
Influenza (Infections and infestations) | 1 | 1
Streptococcal bacteraemia (Infections and infestations) | 2 | 0
Urosepsis (Infections and infestations) | 2 | 0
Abdominal wall abscess (Infections and infestations) | 1 | 0
Abscess (Infections and infestations) | 1 | 0
Abscess neck (Infections and infestations) | 1 | 0
Arteriosclerotic gangrene (Infections and infestations) | 0 | 1
Arteriovenous graft site abscess (Infections and infestations) | 1 | 0
Arthritis infective (Infections and infestations) | 1 | 0
Bacterial disease carrier (Infections and infestations) | 1 | 0
Bronchitis pneumococcal (Infections and infestations) | 1 | 0
Bronchitis viral (Infections and infestations) | 0 | 1
Campylobacter intestinal infection (Infections and infestations) | 1 | 0
Candida sepsis (Infections and infestations) | 0 | 1
Central line infection (Infections and infestations) | 1 | 0
Chest wall abscess (Infections and infestations) | 0 | 1
Clostridial infection (Infections and infestations) | 0 | 1
Emphysematous cystitis (Infections and infestations) | 1 | 0
Empyema (Infections and infestations) | 0 | 1
Endocarditis (Infections and infestations) | 1 | 0
Enterococcal sepsis (Infections and infestations) | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Genital abscess (Infections and infestations) | 0 | 1
Groin abscess (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Intervertebral discitis (Infections and infestations) | 1 | 0
Klebsiella bacteraemia (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Necrotising fasciitis (Infections and infestations) | 1 | 0
Neurosyphilis (Infections and infestations) | 1 | 0
Osteomyelitis chronic (Infections and infestations) | 1 | 0
Paronychia (Infections and infestations) | 1 | 0
Pelvic abscess (Infections and infestations) | 1 | 0
Pleural infection bacterial (Infections and infestations) | 0 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 0
Pneumonia pneumococcal (Infections and infestations) | 0 | 1
Pneumonia primary atypical (Infections and infestations) | 1 | 0
Pneumonia staphylococcal (Infections and infestations) | 0 | 1
Post procedural sepsis (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 1 | 0
Pseudomonal bacteraemia (Infections and infestations) | 1 | 0
Psoas abscess (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Sepsis syndrome (Infections and infestations) | 0 | 1
Septic embolus (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Tracheobronchitis (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 0 | 1
Wound infection bacterial (Infections and infestations) | 0 | 1
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 6 | 8
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 6 | 5
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 6 | 2
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 4 | 2
Femur fracture (Injury, poisoning and procedural complications) | 3 | 2
Hip fracture (Injury, poisoning and procedural complications) | 3 | 2
Vascular graft complication (Injury, poisoning and procedural complications) | 1 | 4
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1 | 3
Arteriovenous fistula aneurysm (Injury, poisoning and procedural complications) | 3 | 0
Arteriovenous graft aneurysm (Injury, poisoning and procedural complications) | 1 | 2
Fall (Injury, poisoning and procedural complications) | 2 | 1
Arteriovenous graft site haemorrhage (Injury, poisoning and procedural complications) | 0 | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 2
Lower limb fracture (Injury, poisoning and procedural complications) | 2 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 2 | 0
Procedural hypotension (Injury, poisoning and procedural complications) | 1 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 1
Back injury (Injury, poisoning and procedural complications) | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Contrast media reaction (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Drug toxicity (Injury, poisoning and procedural complications) | 1 | 0
Eschar (Injury, poisoning and procedural complications) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 1 | 0
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 1 | 0
Open wound (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 | 0
Postoperative fever (Injury, poisoning and procedural complications) | 1 | 0
Pubic rami fracture (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 1 | 0
Skeletal injury (Injury, poisoning and procedural complications) | 1 | 0
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 1 | 0
Occult blood positive (Investigations) | 2 | 0
Alanine aminotransferase decreased (Investigations) | 1 | 0
Anticoagulation drug level above therapeutic (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 1 | 0
International normalised ratio decreased (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 1 | 0
Oxygen saturation decreased (Investigations) | 1 | 0
Prothrombin time shortened (Investigations) | 1 | 0
Sputum culture positive (Investigations) | 0 | 1
Transaminases increased (Investigations) | 1 | 0
Troponin increased (Investigations) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 21 | 18
Hyperkalaemia (Metabolism and nutrition disorders) | 24 | 15
Hypoglycaemia (Metabolism and nutrition disorders) | 8 | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 7 | 1
Dehydration (Metabolism and nutrition disorders) | 3 | 3
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 3 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 3 | 0
Diabetic foot (Metabolism and nutrition disorders) | 2 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 2 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 1 | 0
Calciphylaxis (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemic unconsciousness (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 1
Connective tissue disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 3
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neurilemmoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Refractory anaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Retroperitoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 8 | 8
Syncope (Nervous system disorders) | 6 | 8
Convulsion (Nervous system disorders) | 12 | 1
Transient ischaemic attack (Nervous system disorders) | 5 | 5
Presyncope (Nervous system disorders) | 4 | 1
Anoxic encephalopathy (Nervous system disorders) | 3 | 0
Headache (Nervous system disorders) | 3 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 2
Aphasia (Nervous system disorders) | 0 | 2
Carotid artery stenosis (Nervous system disorders) | 1 | 1
Cerebral infarction (Nervous system disorders) | 0 | 2
Cerebral ischaemia (Nervous system disorders) | 1 | 1
Depressed level of consciousness (Nervous system disorders) | 1 | 1
Facial palsy (Nervous system disorders) | 2 | 0
Haemorrhagic stroke (Nervous system disorders) | 1 | 1
Metabolic encephalopathy (Nervous system disorders) | 1 | 1
Altered state of consciousness (Nervous system disorders) | 1 | 0
Cervical myelopathy (Nervous system disorders) | 1 | 0
Cervicobrachial syndrome (Nervous system disorders) | 1 | 0
Complex partial seizures (Nervous system disorders) | 0 | 1
Dementia Alzheimer's type (Nervous system disorders) | 1 | 0
Diabetic autonomic neuropathy (Nervous system disorders) | 0 | 1
Embolic stroke (Nervous system disorders) | 0 | 1
Encephalitis (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Hypoglycaemic encephalopathy (Nervous system disorders) | 0 | 1
Ischaemic cerebral infarction (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
Lacunar infarction (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0
Lumbar radiculopathy (Nervous system disorders) | 1 | 0
Myoclonic epilepsy (Nervous system disorders) | 1 | 0
Myoclonus (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Reversible ischaemic neurological deficit (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 1
Spinal cord infarction (Nervous system disorders) | 1 | 0
Status epilepticus (Nervous system disorders) | 1 | 0
Thalamus haemorrhage (Nervous system disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 8 | 8
Delirium (Psychiatric disorders) | 2 | 2
Bipolar disorder (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1
Depression suicidal (Psychiatric disorders) | 1 | 0
Homicidal ideation (Psychiatric disorders) | 1 | 0
Schizophrenia, paranoid type (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Renal failure chronic (Renal and urinary disorders) | 4 | 1
Azotaemia (Renal and urinary disorders) | 3 | 1
Bladder perforation (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Nephrosclerosis (Renal and urinary disorders) | 0 | 1
Obstructive uropathy (Renal and urinary disorders) | 1 | 0
Renal cyst (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Ureteric dilatation (Renal and urinary disorders) | 0 | 1
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 2 | 0
Breast calcifications (Reproductive system and breast disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 16 | 5
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 15 | 5
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 8 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 2
Panniculitis (Skin and subcutaneous tissue disorders) | 2 | 0
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Hypotension (Vascular disorders) | 19 | 7
Hypertension (Vascular disorders) | 12 | 5
Hypertensive crisis (Vascular disorders) | 7 | 7
Peripheral vascular disorder (Vascular disorders) | 4 | 4
Accelerated hypertension (Vascular disorders) | 3 | 1
Peripheral ischaemia (Vascular disorders) | 3 | 1
Steal syndrome (Vascular disorders) | 2 | 2
Deep vein thrombosis (Vascular disorders) | 1 | 2
Vascular pseudoaneurysm (Vascular disorders) | 2 | 1
Arteriosclerosis (Vascular disorders) | 1 | 1
Hypertensive emergency (Vascular disorders) | 1 | 1
Malignant hypertension (Vascular disorders) | 2 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 2 | 0
Vena cava thrombosis (Vascular disorders) | 2 | 0
Arterial disorder (Vascular disorders) | 0 | 1
Arterial occlusive disease (Vascular disorders) | 0 | 1
Essential hypertension (Vascular disorders) | 1 | 0
Femoral arterial stenosis (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 1 | 0
Haemorrhage (Vascular disorders) | 0 | 1
Jugular vein thrombosis (Vascular disorders) | 0 | 1
Varicose vein (Vascular disorders) | 0 | 1
Venous stenosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Peginesatide (N=524) | Epoetin Alfa (N=269)
Diarrhoea (Gastrointestinal disorders) | 98 | 35
Nausea (Gastrointestinal disorders) | 89 | 51
Vomiting (Gastrointestinal disorders) | 86 | 32
Constipation (Gastrointestinal disorders) | 37 | 33
Abdominal pain (Gastrointestinal disorders) | 31 | 20
Abdominal pain upper (Gastrointestinal disorders) | 27 | 13
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 17 | 20
Haemorrhoids (Gastrointestinal disorders) | 7 | 14
Pyrexia (General disorders) | 62 | 39
Oedema peripheral (General disorders) | 45 | 23
Asthenia (General disorders) | 41 | 16
Fatigue (General disorders) | 33 | 20
Pain (General disorders) | 24 | 15
Chills (General disorders) | 20 | 16
Upper respiratory tract infection (Infections and infestations) | 61 | 40
Urinary tract infection (Infections and infestations) | 40 | 26
Nasopharyngitis (Infections and infestations) | 37 | 25
Bronchitis (Infections and infestations) | 35 | 12
Sinusitis (Infections and infestations) | 27 | 13
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 77 | 43
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 42 | 24
Vascular graft complication (Injury, poisoning and procedural complications) | 39 | 24
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 38 | 15
Fall (Injury, poisoning and procedural complications) | 38 | 15
Procedural hypotension (Injury, poisoning and procedural complications) | 33 | 23
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 31 | 7
Hyperkalaemia (Metabolism and nutrition disorders) | 32 | 25
Fluid overload (Metabolism and nutrition disorders) | 20 | 17
Muscle spasms (Musculoskeletal and connective tissue disorders) | 57 | 40
Pain in extremity (Musculoskeletal and connective tissue disorders) | 54 | 32
Back pain (Musculoskeletal and connective tissue disorders) | 51 | 35
Arthralgia (Musculoskeletal and connective tissue disorders) | 49 | 25
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 26 | 20
Headache (Nervous system disorders) | 74 | 40
Dizziness (Nervous system disorders) | 55 | 33
Insomnia (Psychiatric disorders) | 34 | 20
Anxiety (Psychiatric disorders) | 31 | 15
Cough (Respiratory, thoracic and mediastinal disorders) | 101 | 52
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 89 | 51
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 23 | 15
Pruritus (Skin and subcutaneous tissue disorders) | 27 | 16
Hypotension (Vascular disorders) | 49 | 27
Hypertension (Vascular disorders) | 43 | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first publication of the primary safety and efficacy results will include data from all appropriate study sites. Either after the first multicenter publication, or following 36 months after the completion of the study, Investigators are free to publish; such publications may not contain Sponsor Confidential Information and may be subject to Sponsor review 60 days prior to submission for publication.